CLINICAL TRIAL: NCT01654458
Title: A Randomized Controlled Trial of an Online Support Group for Sexual Distress Due to Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other); Tom Baker Cancer Centre (Other); Cross Cancer Institute (Other); Vancouver Coastal Health Research Institute (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OVA-120243; 1009695 (Other: Women's College Hospital Research Ethics Board); 12-0427-CE (Other: University Health Network Research Ethics Board); 216-2012 (Other: Research Ethics Board of Sunnybrook Health Sciences Centre)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Sexual Dysfunctions, Psychological; Uterine Cervical Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female
Keywords: Sexual Dysfunctions, Psychological; Psychotherapy, Group; Genital Neoplasms, Female; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Urogenital Neoplasms; Uterine Cervical Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Uterine Cervical Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female; Endometrial Neoplasms; Fallopian Tube Neoplasms; Urogenital Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Treatment Condition (Experimental): Receives the 12-week GyneGals Support Group within a month of completing the baseline assessment.
  Interventions: Behavioral: GyneGals Support Group
- Waitlist Control Condition (No Intervention): Waitlist control group receives the 12-week GyneGals Support Group only after its involvement in the study has ended, as a courtesy.

INTERVENTIONS:
Behavioral: GyneGals Support Group — 12-week online (i.e. Internet-based), professionally-facilitated support group
  Arms: Immediate Treatment Condition

SUMMARY:
There is a high prevalence of sexual and body image problems among women treated for gynecologic cancer, which can lead to considerable distress. Given the sensitive and highly personal nature of these problems, women are often reluctant to speak to their doctors about these concerns and have few resources for support and information. The research team will conduct a prospective randomized controlled trail (RCT) to test the benefits of "GyneGals," a 12-week online (i.e. Internet-based) support group intervention for women who are sexually distressed due to gynecologic cancer and its treatment.

The primary aim of this study is to determine whether a professionally-facilitated, information-rich, online support group is beneficial for women who are sexually distressed due to gynecologic cancer and the side effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Received surgical, radiation or chemotherapy treatments for any gynecologic cancer
* Not receiving active treatment
* Currently disease-free for a minimum of 3 months
* No more than 5 years post-diagnosis
* Distressed due to psychosexual concerns related to cancer
* Willing to discuss psychosexual concerns
* 18 years or older
* Has access to a computer and the Internet
* Speaks, reads, and writes in English
* Provides informed consent

Exclusion Criteria:

* Acutely suicidal (i.e., actively suicidal within the previous 3 months)
* Has a major psychiatric illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2012-07; Primary Completion 2018-01-19 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Psychosexual distress, as measured by the Revised Female Sexual Distress Scale (FSDS-R). | 9 months
  13-item self-report scale that measures sexually-related distress in women.

SECONDARY OUTCOMES:
Sexual function, as measured by the Sexual Function Questionnaire (SFQ). | 9 months (at months 1, 5, and 9)
  25-item measure developed for cancer patients and can be completed by women regardless of sexual orientation or whether they have a partner.
Body image, as measured by the Sexual Adjustment and Body Image Scale - Gynecologic Cancer (SABIS-G). | 9 months (at months 1, 5, and 9)
  Consists of two independent scales designed to assess changes in sexuality and body image before and after diagnosis.
Depression and anxiety symptoms, as measured by the Hospital Anxiety and Depression Scale (HADS). | 9 months (at months 1, 5, and 9)
  14-item self-report questionnaire for detecting depression and anxiety in a hospital outpatient setting.
Relationship satisfaction, as measured by the Relationship Assessment Scale (RAS). | 9 months (at months 1, 5, and 9)
  7-item measure assessing satisfaction with an individual's romantic relationship.
Perceived social support, as measured by MOS Social Support Survey (MOS-SS). | 9 months (at months 1, 5, and 9)
  19 items and assesses emotional/informational support, tangible support, affectionate support, and positive social interaction, as well as providing an overall functional support index.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine C. Classen, PhD, Principal Investigator — Women's College Hospital
Locations (7):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network (Princess Margaret Hospital), Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

REFERENCES:
- [Background] Classen CC, Chivers ML, Urowitz S, Barbera L, Wiljer D, O'Rinn S, Ferguson SE. Psychosexual distress in women with gynecologic cancer: a feasibility study of an online support group. Psychooncology. 2013 Apr;22(4):930-5. doi: 10.1002/pon.3058. Epub 2012 Feb 28. PMID 22374732
- [Background] Wiljer D, Urowitz S, Barbera L, Chivers ML, Quartey NK, Ferguson SE, To M, Classen CC. A qualitative study of an internet-based support group for women with sexual distress due to gynecologic cancer. J Cancer Educ. 2011 Sep;26(3):451-8. doi: 10.1007/s13187-011-0215-1. PMID 21594587
- [Background] Classen CC, Drozd A, Brotto LA, Barbera L, Carter J, Chivers ML, Koval J, Robinson JW, Urowtiz S, Wiljer D, & Ferguson SE. Protocol of a randomized controlled trial of an online support group for sexual distress due to gynecologic caner. Journal of Clinical Trials 5(4), 2015. DOI: 10.4172/2167-0870.1000234